CLINICAL TRIAL: NCT03250078
Title: A Pancreatic Cancer Screening Study in Hereditary High Risk Individuals
Status: Recruiting | Type: Observational
Sponsor: Nuvance Health (Other)
Responsible Party: Principal Investigator, Richard Frank, Director, Cancer Research, Nuvance Health
Other Study IDs: 16-17
Record Dates: First submitted 2016-11-16; First posted 2017-08-15 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Pancreatic Neoplasms
Keywords: Pancreas; Cancer; MRI; BRCA; Early Detection; Genetics; ATM; PALB2; Lynch; CDKN2A
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FAMILIAL PANCREATIC CANCER and/or GENE MUTATION: An inherited genetic syndrome associated with Pancreatic Cancer and/or with a strong family history of Pancreatic Cancer.
  Interventions: Diagnostic Test: MRI/MRCP

INTERVENTIONS:
Diagnostic Test: MRI/MRCP — An MRI/MRCP plus IV gadolinium contrast with high resolution imaging of the pancreas will be performed annually

SUMMARY:
The main goal of this study is to screen and detect pancreatic cancer and precursor lesions in individuals with a strong family history or genetic predisposition to pancreatic cancer. Magnetic Resonance Imaging and Magnetic cholangiopancreatography (MRI/MRCP) will be utilized to screen for early stage pancreatic cancer or precursor lesions. Participants will be asked to donate a blood sample at specific intervals for the creation of a bio-bank necessary for the development of a blood based screening test for Pancreatic Cancer.

DETAILED DESCRIPTION:
Individuals 50 years of age and older who have a family history of pancreatic cancer will be recruited through the offices of primary care physicians and endocrinologists. Those meeting initial criteria will meet with a research APRN and will undergo a secondary screen to determine eligibility. Individuals enrolled in the study will undergo a five-minute psychological survey and donation of a blood sample for bio-bank analysis every 6 months for 3 years. MRI will be performed annually for 3 years (4 in total). Any abnormalities on MRI will be reviewed by a multi-disciplinary tumor board and discussed with the participant. The costs of MRI will be covered by the study.

ELIGIBILITY:
Registration-Inclusion Criteria for FAMILIAL PANCREATIC CANCER (FPC) and those with a BRCA1, BRCA2, LYNCH SYNDROME, ATM, PALB2, CDKN2A, or related gene mutation (one of the following is required for questions 1-3)

1. For FPC: The individual has at least 2 first-degree relatives (FDR) with PC.
2. For FPC: The individual has at least 3 first-, second-, or third-degree relatives with PC with at least 1 PC in a FDR.
3. The individual is a known mutation carrier of BRCA1, BRCA2, MLH1, MSH2, MSH6, or PMS2, ATM, PALB2, CDKN2A, or similar high-risk gene mutation and has at least 1 first- or second-degree relative with PC.
4. The individual is at least 50 years old or 10 years younger than the youngest relative with PC.
5. ECOG Performance Status of 0-1.
6. No known contraindications to MRI examination or gadolinium contrast.
7. Willing to undergo MRI and screening for metal implants or metal injury.
8. Estimated GFR >29 mL/min
9. Ability to provide informed consent.
10. Willing to return to study site for all study assessments.

Registration-Exclusion Criteria:

1. Prior history of pancreatic cancer.
2. Presence of metastatic cancer or cancer requiring adjuvant chemotherapy within the past 5 years.
3. Received chemotherapy within the past 6 months. (Hormonal therapy is allowable if the disease free interval is at least 5 years).
4. Hereditary pancreatitis.
5. eGFR < 30 mL/min
6. Contraindication to MRI examination or gadolinium contrast.
7. Pregnant or nursing women.
8. Co-morbid illnesses or other concurrent disease which, in the judgment of the clinicians obtaining informed consent, would make the participant inappropriate for entry into this study.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50-90 years of age. Strong family history of pancreatic cancer/ known genetic mutation
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-11; Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Early Stage Pancreatic Cancer or Precursor Lesions | Through study completion, up to 3 years
  Incidence of Pancreatic Cancer or precursor lesions within a population of individuals with a strong family history of pancreatic cancer or known genetic mutation compared to the expected incidence in the general population.

SECONDARY OUTCOMES:
Serial Pancreatic MRI Screening | Through study completion, up to 3 years
  Utility of MRI as a screening tool for Pancreatic Cancer in the study population.
Serum Bio-bank | Through study completion, up to 3 years
  Banking serum from participants to isolate circulating exosomes and circulating tumor DNA.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Frank, MD, Principal Investigator — Nuvance Health
Locations (1):
- Nuvance Health, Norwalk, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed on an individual basis post submission. Requestors may be required to sign a data access agreement.

REFERENCES:
- [Derived] Kandiah J, Lo T, Jin D, Melchior L, Krebs TL, Anand N, Ingram S, Krumholtz P, Pandya D, Trinidad A, Dong XE, Seshadri R, Bauman J, Lee R, Frank RC. A Community-Based Pancreatic Cancer Screening Study in High-Risk Individuals: Preliminary Efficacy and Safety Results. Clin Transl Gastroenterol. 2022 Aug 1;13(8):e00516. doi: 10.14309/ctg.0000000000000516. Epub 2022 Jul 20. PMID 35854467
- See also: An overview pancreatic cancer research at Nuvance Health — https://www.nuvancehealth.org/about-us/research-and-innovation/cancer-research/pancreatic-cancer-research